CLINICAL TRIAL: NCT04616196
Title: A Phase 1b/2, Open-label, Multicenter, Dose Escalation and Dose Expansion Study of NKTR-255 Monotherapy or in Combination With Cetuximab as a Salvage Regimen for Solid Tumors
Brief Title: Study of NKTR 255 in Combination With Cetuximab in Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-255-03
Record Dates: First submitted 2020-10-30; First posted 2020-11-04 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Colorectal Cancer
Keywords: HNSCC; Head and Neck Squamous Cell Carcinoma; CRC; Colorectal Cancer; NKTR-255; Cetuximab; Erbitux®
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms | interventions — NKTR-255; Cetuximab

STUDY DESIGN:
Intervention Model Description: Phase 1: Dose escalation cohorts will be sequential
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation of NKTR-255 with Cetuximab (Experimental): Establish RP2D, of NKTR-255 with cetuximab.
  Interventions: Drug: NKTR-255; Drug: Cetuximab

INTERVENTIONS:
Drug: NKTR-255 — NKTR-255 IV every 21 days
Drug: Cetuximab — Cetuximab will be given at specified doses on specified days
  Other Names: Erbitux®

SUMMARY:
This is a Phase 1b/2, open-label multicenter study evaluating NKTR-255 as a monotherapy and together with cetuximab in patients with head and neck squamous cell carcinoma (HNSCC) and colorectal carcinoma (CRC).

DETAILED DESCRIPTION:
NKTR-255 is a cytokine that is designed to regulate T and natural killer cell activation, proliferation and promote their anti-tumor effects.

In the dose escalation (Phase 1/b) phase patients with HNSCC or CRC will be treated with ascending doses of NKTR-255 in combination with cetuximab, until the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) is reached.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of a locally advanced or metastatic HNSCC or CRC.
* Life expectancy > 12 weeks as determined by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Measurable disease per RECIST 1.1.

HNSCC:

* Progression on any first or second line platinum-based chemotherapy and/or anti-PD-1 or programmed death-ligand 1 antibody.

CRC:

* Patients must have received or were intolerant to at least 2 prior cancer therapy regimens administered for metastatic disease.

Key Exclusion Criteria:

* Use of an investigational agent or an investigational device within 28 days before administration of first dose of study drug(s)
* Prior surgery or radiotherapy within 14 days of initiating study drug(s)
* Evidence of clinically significant interstitial lung disease or active, noninfectious pneumonitis; active infection requiring systemic therapy within 7 days prior to dosing
* Patients who have been previously treated with IL-2 or IL-15
* Known Grade 3 or 4 hypersensitivity reaction to cetuximab, history of allergy to red meat or tick bites, or history of positive test results for immunoglobulin E antibodies against cetuximab
* Patients who have an active, known, or suspected autoimmune disease

NOTE: Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (6):
- United States (6):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - START Center for Cancer Care, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Phase 1 portion of the study was completed. The Phase 2 cohort enrollment was not initiated.
Groups:
- Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab; Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab; Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab; Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab: Establish RP2D, of NKTR-255 with cetuximab.
  NKTR-255: NKTR-255 IV every 21 days
  Cetuximab: Cetuximab will be given at specified doses on specified days
Period: Overall Study
Arm/Group | Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab
Started (This is based on the Enrolled Population, patients who received at least one dose (or partial dose) of cetuximab or NKTR-255. However, only 23 were dosed with NKTR-255 (7 in Level 1, 7 in Level 2, 6 in Level 3, 3 in Level 4) and are included in the Safety Population analysis used for the remainder of results data.) | 8 | 8 | 6 | 3
Number of Participants Who Were Included in the "Safety Population" Analysis. | 7 | 7 | 6 | 3
Completed | 0 | 1 | 0 | 0
Not Completed | 8 | 7 | 6 | 3
Not completed — Progressive Disease | 3 | 0 | 4 | 1
Not completed — Death | 2 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Sponsor request | 2 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Only 23 participants were dosed with NKTR-255 (7 in Level 1, 7 in Level 2, 6 in Level 3, 3 in Level 4) and are included in the Safety Population analysis used for the remainder of results data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab | Total
Number analyzed (Participants) | 7 | 7 | 6 | 3 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (7.3) | 56.9 (11.44) | 60.7 (18.02) | 59.0 (11.00) | 59.3 (11.75)
Age, Customized [Number; unit: participants]
  <65 | 5 | 4 | 3 | 2 | 14
  >=65 and <75 | 2 | 3 | 2 | 1 | 8
  >=75 and <85 | 0 | 0 | 1 | 0 | 1
  >=85 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 1 | 6
  Male | 7 | 5 | 3 | 2 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 5 | 6 | 4 | 3 | 18
  Not Reported | 1 | 0 | 0 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 4 | 5 | 5 | 1 | 15
  Unknown | 1 | 0 | 1 | 0 | 2
  Not Reported | 1 | 1 | 0 | 1 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Participants must meet the ECOG Performance status of 0 or 1 criteria for enrollment in the study.
  ECOG Performance Status of 0 = Able to carry out all normal activities without restriction. ECOG Performance Status of 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature.
  Participants
    ECOG PS 0 | 2 | 4 | 3 | 1 | 10
    ECOG PS 1 | 5 | 3 | 3 | 2 | 13
Height [Mean (Standard Deviation); unit: centimeter] — Population: The number analyzed for height is less than the overall number of baseline participants, since there was missing patient data.
  centimeter
    number analyzed (Participants) | 6 | 7 | 6 | 2 | 21
    (all) | 176.69 (6.370) | 171.78 (7.202) | 167.90 (14.675) | 168.54 (3.062) | 171.76 (9.635)
Weight [Mean (Standard Deviation); unit: kg] | 91.77 (14.415) | 84.20 (14.359) | 87.46 (44.884) | 70.98 (17.727) | 85.63 (25.341)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: The number analyzed for BMI is less than the overall number of baseline participants, since there was missing patient data.
  kg/m^2
    number analyzed (Participants) | 6 | 7 | 6 | 2 | 21
    (all) | 30.13 (4.227) | 28.89 (6.997) | 29.98 (10.569) | 22.00 (4.414) | 28.90 (7.323)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE) of NKTR-255 in Combination With Cetuximab in R/R HNSCC or CRC for Phase 1b Dose Escalation
Description: Safety and tolerability of NKTR-255 in combination with cetuximab as evaluated by dose limiting toxicities, incidence of drug-related Adverse Events (AEs), SAEs, and AEs leading to discontinuation, deaths, and clinical laboratory abnormalities per CTCAE 5.0
Time Frame: 60 days after the last dose of study treatment, up to an average of 6 months.
Population: DLTs were assessed using the DLT Population, which only included patients who received at least 1 dose of the combination treatment of NKTR-255 and cetuximab and who completed the DLT observation period or discontinued from the study treatment due to a DLT, where DLT window was 21 days since the first dose of NKTR-255. The other rows were assessed using the Safety Population, patients who received at least 1 dose (or partial dose) of NKTR-255.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab; Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab; Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab; Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab: NKTR-255: NKTR-255 IV every 21 days
  Cetuximab: Cetuximab will be given at specified doses on specified days
Arm/Group | Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab
Number analyzed (Participants) | 7 | 7 | 6 | 3
Participants
  Patients with dose limiting toxicities (DLTs): Infusion related reaction: number analyzed (Participants) | 6 | 6 | 6 | 2
  Patients with dose limiting toxicities (DLTs): Infusion related reaction | 0 | 1 | 0 | 0
  Patients With at Least one TEAE | 7 | 7 | 6 | 2
  Patients With at Least one TEAE Related to NKTR-255 | 5 | 7 | 5 | 2
  Patients With at Least one Serious TEAE | 2 | 2 | 5 | 1
  Patients With at Least one Serious TEAE Related to NKTR-255 | 0 | 1 | 0 | 1
  Patients With at Least one TEAE Leading to Death | 0 | 0 | 0 | 0
  Patients With at Least one TEAE Related to NKTR-255 Leading to Death | 0 | 0 | 0 | 0
  Patients With at Least one TEAE Leading to NKTR-255 Discontinuation | 0 | 2 | 0 | 0
  Patients With at Least one TEAE Leading to NKTR-255 Delay, Reduction, or Interruption | 2 | 0 | 2 | 0

2. Primary Outcome: The Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of NKTR-255 in Combination With Cetuximab in R/R HNSCC or CRC for Phase 1b Dose Escalation
Description: To define the MTD and/or RP2D of NKTR-255 in combination with cetuximab in R/R HNSCC or CRC for Phase 1b Dose Escalation
Time Frame: Up to 21 days
Measure: Number; unit: µg/kg
Arm/Group | Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab
Number analyzed (Participants) | 7 | 7 | 6 | 3
µg/kg | NA — MTD was not established. There were no dose limiting toxicity in the highest dose of 6 µg/kg and above, therefore there was no MTD. | NA — MTD was not established. There were no dose limiting toxicity in the highest dose of 6 µg/kg and above, therefore there was no MTD. | NA — MTD was not established. There were no dose limiting toxicity in the highest dose of 6 µg/kg and above, therefore there was no MTD. | NA — MTD was not established. There were no dose limiting toxicity in the highest dose of 6 µg/kg and above, therefore there was no MTD.

ADVERSE EVENTS:
Time Frame: Through study completion, up to 6 months.
Description: Adverse events were collected through regular investigator assessments and regular laboratory testing.
Arm/Group | Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab | Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab
All-Cause Mortality (participants affected / at risk) | 2/8 | 4/8 | 1/6 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/7 | 5/6 | 1/3
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 6/6 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab (N=7) | Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab (N=7) | Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab (N=6) | Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab (N=3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation of NKTR-255 Level 1 (1.5 µg/kg) With Cetuximab (N=7) | Dose Escalation of NKTR-255 Level 2 (3.0 µg/kg) With Cetuximab (N=7) | Dose Escalation of NKTR-255 Level 3 (4.5 µg/kg) With Cetuximab (N=6) | Dose Escalation of NKTR-255 Level 4 (6.0 µg/kg) With Cetuximab (N=3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 4 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Chills (General disorders) | 1 | 1 | 2 | 1
Fatigue (General disorders) | 1 | 2 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Ascites (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 6 | 1 | 0
Paronychia (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pyuria (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT04616196/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT04616196/SAP_001.pdf